CLINICAL TRIAL: NCT03080987
Title: A 2-Part Study to Assess the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Pharmacodynamics of JNJ-64179375 in Healthy Japanese Subjects
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Pharmacodynamics of JNJ-64179375 in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108306; 2016-004785-25 (EudraCT Number); 64179375EDI1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-03-10; First posted 2017-03-15 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part 1: Cohort 1 (0.3 mg/kg of JNJ-64179375 or Placebo) (Experimental): Participants will receive a single 0.3 milligram per kilogram (mg/kg) intravenous (IV) dose of JNJ-64179375 or matching Placebo on Day 1.
  Interventions: Drug: JNJ-64179375 0.3 mg/kg; Other: Placebo
- Part 1: Cohort 2 (1.0 mg/kg of JNJ-64179375 or Placebo) (Experimental): Participants will receive a single 1.0 mg/kg IV dose of JNJ-64179375 or matching Placebo on Day 1.
  Interventions: Drug: JNJ-64179375 1.0 mg/kg; Other: Placebo
- Part 1: Cohort 3 (2.5 mg/kg of JNJ-64179375 or Placebo) (Experimental): Participants will receive a single 2.5 mg/kg IV dose of JNJ-64179375 or matching Placebo on Day 1.
  Interventions: Drug: JNJ-64179375 2.5 mg/kg; Other: Placebo
- Part 1: Optional Cohort 1 (JNJ-64179375 or Placebo) (Experimental): Participants will receive a single IV dose of JNJ-64179375 (dose to be determined) or matching Placebo on Day 1.
  Interventions: Other: Placebo; Drug: JNJ-64179375 (Dose to be Determined)
- Part 1: Optional Cohort 2 (JNJ-64179375 or Placebo) (Experimental): Participants will receive a single IV dose of JNJ-64179375 (dose to be determined) or matching Placebo on Day 1.
  Interventions: Other: Placebo; Drug: JNJ-64179375 (Dose to be Determined)
- Part 2: SC Cohort (1.0 mg/kg of JNJ-64179375 or Placebo) (Experimental): Participants will receive a single subcutaneous (SC) dose of 1.0 mg/kg or highest tolerable dose if less than 1.0 mg/kg of JNJ-64179375 or matching Placebo on Day 1.
  Interventions: Drug: JNJ-64179375 1.0 mg/kg; Other: Placebo

INTERVENTIONS:
Drug: JNJ-64179375 0.3 mg/kg — JNJ-64179375 0.3 milligram per kilogram (mg/kg) intravenous (IV) infusion on Day 1.
  Arms: Part 1: Cohort 1 (0.3 mg/kg of JNJ-64179375 or Placebo)
Drug: JNJ-64179375 1.0 mg/kg — JNJ-64179375 1.0 mg/kg on Day 1 administered as IV infusion (for Part 1) and SC injection (for Part 2).
  Arms: Part 1: Cohort 2 (1.0 mg/kg of JNJ-64179375 or Placebo); Part 2: SC Cohort (1.0 mg/kg of JNJ-64179375 or Placebo)
Drug: JNJ-64179375 2.5 mg/kg — JNJ-64179375 2.5 mg/kg IV infusion on Day 1.
  Arms: Part 1: Cohort 3 (2.5 mg/kg of JNJ-64179375 or Placebo)
Other: Placebo — Matching placebo on Day 1 administered as IV infusion (for Part 1) and SC injection (for Part 2).
Drug: JNJ-64179375 (Dose to be Determined) — JNJ-64179375 IV infusion (Dose to be determined).
  Arms: Part 1: Optional Cohort 1 (JNJ-64179375 or Placebo); Part 1: Optional Cohort 2 (JNJ-64179375 or Placebo)

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of JNJ-64179375 in Part 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Must have been born in Japan of Japanese parents and maternal and paternal Japanese grandparents
* Body mass index (weight kg/m^2) between 18 and 27 kilogram per square meter (kg/m^2) (inclusive), and body weight greater than 50 kg but less than 100 kg
* Generally in good health on the basis of physical examinations, medical history, vital signs, laboratory tests, electrocardiograms (ECGs) and cardiac telemetry performed at Screening and/or prior to administration of the initial dose of study drug
* Must sign an informed consent form (ICF) indicating that he understands the purpose of, and procedures required for, the study and is willing to participate in the study

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, bleeding or thrombotic disorders (including any personal or family history of abnormal bleeding as assessed by a detailed bleeding history or blood dyscrasias), or with an underlying coagulopathy that may lead to a clinically relevant bleeding risk, autoimmune disease, lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the subject or that could interfere with the interpretation of the study results
* Acute illness, including an upper respiratory infection (with or without fever), within 7 days prior to study drug administration or have had a major illness or hospitalization within 1 month prior to study drug administration
* Clinically significant abnormal physical exam at Screening or Day -1
* Clinically significant abnormal vital signs at Screening, Day -1, or Day 1 (predose) as determined by the investigator or appropriate designee
* Clinically significant abnormal cardiac telemetry, or ECG at Screening, Day -1, or Day 1 (predose) as determined by the investigator or appropriate designee

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Up to Day 113
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Part 2: Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Up to Day 113
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

SECONDARY OUTCOMES:
Part 1 and 2: Maximum Observed Plasma Concentration (Cmax) of JNJ-64179375 | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113 post-dose
  Cmax is the maximum observed plasma concentration.
Part 1 and 2: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) of JNJ-64179375 | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113 post-dose
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Part 1 and 2: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of JNJ-64179375 | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113 post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time.
Part 1: Total Systemic Clearance (CL) of JNJ-64179375 | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113 post-dose
  CL is defined as total systemic clearance after intravenous administration of JNJ-64179375.
Part 1: Apparent Volume of Distribution at Terminal Phase After Intravenous Administration (Vz) of JNJ-64179375 | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113 post-dose
  Vz is defined as the Apparent volume of distribution at terminal phase after intravenous administration.
Part 1 and 2: Terminal Half-Life (t1/2) of JNJ-64179375 | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113 post-dose
  Half-life is the time measured for the plasma concentration of drug to decrease by one half.
Part 2: Total Systemic Clearance Over Bioavailability After Subcutaneous (SC) Administration (CL/F) of JNJ-64179375 post-dose | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113 post-dose
  CL/F is defined as total systemic clearance over bioavailability after SC administration.
Part 2: Apparent Volume of Distribution at Terminal Phase Over Bioavailability After Subcutaneous Administration (Vz/F) of JNJ-64179375 | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113 post-dose
  (Vz/F) is defined as Apparent Volume of distribution at terminal phase over bioavailability after SC administration of JNJ-64179375.
Part 2: Absolute Bioavailability (F) After Subcutaneous Administration of JNJ-64179375 | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113 post-dose
  F is defined as absolute bioavailability after SC administration of JNJ-64179375.
Part 1 and 2: Immunogenicity of JNJ-64179375 | Predose, Day 7, 14, 29, 57, 85 and 113 post-dose
  Plasma samples will be collected and screened for antibodies binding to JNJ-64179375 and the titer of confirmed positive samples will be reported.
Part 1 and 2: Pharmacodynamic Effect of JNJ-64179375 as Assessed by Change in Thrombin Time (TT) | Predose, Day 1, 2, 4, 7, 14, 29, 57 and 113 post-dose
  The pharmacodynamic effect of JNJ-64179375 on coagulation parameters will be assessed by measuring the change in thrombin time (TT).
Part 1 and 2: Pharmacodynamic Effect of JNJ-64179375 as Assessed by Change in Prothrombin Time (PT) | Predose, Day 1, 2, 4, 7, 14, 29, 57 and 113 post-dose
  The pharmacodynamic effect of JNJ-64179375 on coagulation parameters will be assessed by measuring the change in prothrombin time (PT).
Part 1 and 2: Pharmacodynamic Effect of JNJ-64179375 as Assessed by Change in Activated Partial Thromboplastin time (aPTT) | Predose, Day 1, 2, 4, 7, 14, 29, 57 and 113 post-dose
  The pharmacodynamic effect of JNJ-64179375 on coagulation parameters will be assessed by measuring the change in activated partial thromboplastin time (aPTT).
Part 1 and 2: Pharmacodynamic Effect of JNJ-64179375 as Assessed by Change in Ecarin Clotting time (ECT) | Predose, Day 1, 2, 4, and 14 post-dose
  The pharmacodynamic effect of JNJ-64179375 on coagulation parameters will be assessed by measuring the change in Ecarin Clotting time (ECT).
Part 1 and 2: Pharmacodynamic Effect of JNJ-64179375 on Platelet Function | Predose, Days 1 and 14 post-dose
  Platelet function will be assessed by measuring platelet activation and aggregation in response to thrombin and other agonists and with the platelet function analyzer (PFA)100.
Part 1 and 2: Pharmacodynamic Effect of JNJ-64179375 as Assessed by Thrombin Generation Assay (TGA) | Predose, Day 1 and 14 post-dose
  The TGA is based on the premise that measurements of thrombin generation are indicative of the overall coagulating capacity of the individual.
Part 1 and 2: Pharmacodynamic Effect of JNJ-64179375 as Assessed by D-dimer | Predose, Day 1 and 14 post-dose
  The D-dimer assay is an enzyme immunoassay procedure for the quantitative determination of D-dimer.
Part 1 and 2: Pharmacodynamic Effect of JNJ-64179375 as Assessed by Change in International Normalized Ratio (INR) | Predose, Day 1, 2,4, 7, 14, 29, 57 and 113 post-dose
  The pharmacodynamic effect of JNJ-64179375 on coagulation parameters will be assessed by measuring the change in international normalized ratio (INR).
Part 2: Time to Maximum Observed Plasma Concentration (Tmax) After Subcutaneous Administration of JNJ-64179375 | Predose, Day 1, 2,4, 7, 10, 14, 22, 29,43, 57, 85 and 113 post-dose
  The Tmax is defined as actual sampling time to reach maximum observed plasma concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- Souseikai Hakata Clinic, Fukuoka, Japan
- Hammersmith Medicines Research Ltd, London, United Kingdom